CLINICAL TRIAL: NCT04780113
Title: Evaluation of Evolution of Perceived Stress in General Practice Residents of Rouen and Caen During COVID-19 Sanitary Crisis
Brief Title: Evolution of Perceived Stress in General Practice Residents During COVID-19 Sanitary Crisis
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Eure-Seine (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03283-36; CHES N°20/01 (Other: CH Eure-Seine)
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the last several years, distress among healthcare professionals is well described, and general practice residents are also affected. Because of COVID-19 sanitary crisis, stress factors are increased, and that may cause anxiety, exhaustion, psychic distress, depression, addictions, or post traumatic stress.

DETAILED DESCRIPTION:
This prospective non-interventional study aims to evaluate via two questionnaires the evolution of perceived stress in general practice residents of two centres in France, Rouen and Caen. The two questionnaires contain the Perceived Stress Scale, as well as items regarding socio-demographic data and stress factors. The first questionnaire is to be distributed during the epidemic COVID-19 wave and the second questionnaire at the end of the epidemic COVID-19 wave.

ELIGIBILITY:
Inclusion Criteria:

* Being a general practice resident in Rouen or Caen
* Participant informed and non-objection of him/her

Exclusion Criteria:

* Being on maternity leave or not working during the period concerned with the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants being general practice residents in Caen or Rouen
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Evolution of perceived stress during the epidemic wave of COVID19 vs. at the end of the epidemic wave of COVID19 | maximum 6 months, according to the evolution of the epidemic
  The perceived stress will be evaluated using the Perceived Stress Scale. This scale contains 10 items, with scores ranging from 0 to 40, with higher scores meaning a higher level of stress.

SECONDARY OUTCOMES:
Description of general characteristics of residents and their feelings and experiences with the sanitary crisis | maximum 6 months, according to the evolution of the epidemic
  This include socio-demographic characteristics, work-related information and potential stress factors
Assessment of residents' profile stress according to their socio-demographic and working characteristics | maximum 6 months, according to the evolution of the epidemic
  Identification of stress factors among residents

CONTACTS AND LOCATIONS:
Overall Officials: Ségolène Guillemette, MD, Principal Investigator — General Practice Physician
Locations (1):
- CH Eure-Seine, Évreux, France